CLINICAL TRIAL: NCT00447473
Title: Phase II Trial to Assess the Activity of Ketoconazole and Mitoxantrone Plus GM-CSF in Patients With Progressive Hormone Refractory Prostate Cancer
Brief Title: Trial of GM-CSF Given in Combination With Ketoconazole and Mitoxantrone in Patients With Progressive Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMRI IRB#0106-0010; PC-Keto-Mito.2006 (Other: Principal Investigator)
Record Dates: First submitted 2007-03-12; First posted 2007-03-14 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Prostatic Neoplasms
Keywords: Prostate Cancer; progressive hormone refractory prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Granulocyte-Macrophage Colony-Stimulating Factor; sargramostim; Ketoconazole; Mitoxantrone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Other): GM-CSF given in combination with ketoconazole and mitoxantrone in patients with progressive prostate cancer despite androgen deprivation and prior taxane containing chemotherapy
  Interventions: Drug: GM-CSF; Drug: Ketoconazole; Drug: Mitoxantrone

INTERVENTIONS:
Drug: GM-CSF — GM-CSF will be administered as a subcutaneous injection at a dose of 250mcg/m2/d (maximum 500 mcg) on weeks 2 and 3 each 21 day cycle (total of 14 days).
  Other Names: Leukine
Drug: Ketoconazole — Ketoconazole will be administered daily at a dose of 400 mg po tid (either 1 hour before or 2 hours after meals), ascorbic acid 250 mg po tid (given with ketoconazole) and replacement doses of hydrocortisone (20 mg po in the morning and 10 mg po in the evening).
  Other Names: Nizoral, Extina, Xolegel, Kuric
Drug: Mitoxantrone — Mitoxantrone will be given at dose of 12 mg/m2 every 3 weeks, up to a maximum cumulative dose of 140 mg/m2
  Other Names: Novantrone, Mitoxantrone

SUMMARY:
This trial represents an attempt to offer second line immunotherapy plus chemotherapy to patients who have failed prior taxane base therapy.

DETAILED DESCRIPTION:
Prostate cancer is the second leading cause of cancer death in American men. Hormonal ablation, in the form of medical or surgical castration is the cornerstone of management for metastatic prostate cancer however, treatment options for a patient in whom androgen ablation fails are limited. Second-line hormonal agents are generally associated with low response rates and no documented survival benefit.

A variety of taxane-based regimens have been tested in hormone refractory prostate cancer, yielding response rates between 38% - 69%. As responses to taxane-based regimens have appeared to exceed those typically associated with mitoxantrone plus prednisone, taxane-based therapy has been widely used in the community, typically as first line therapy. Second line therapy, which are non-taxane based and have comparable activities do not exist.

This study builds on experience in drug development for advanced prostate cancer demonstrating the following:

1. Ketoconazole produces serologic and objective clinical responses in over 50% of patients with disease progression on oral antiandrogen.
2. GM-CSF, as a potent stimulator of dendritic cells, has demonstrated clinical activity in prostate cancer.
3. GM-CSF is well tolerated in patients with prostate cancer. The addition of GM-CSF to antitumor therapy may augment the T cell response to apoptotic tumor cells and therefore may improve the clinical benefit produced by such agents.
4. The addition of mitoxantrone with ketoconazole demonstrated improved clinical benefit relative to the published data with each single agent.

The importance of this trial in the broader context of clinical research for prostate cancer is twofold: One, it represents an attempt to offer second line immunotherapy plus chemotherapy to patients who have failed prior frontline taxane based therapy. Two, this is the first trial to assess the combination of GM-CSF plus ketoconazole and mitoxantrone.

ELIGIBILITY:
* Histologically confirmed adenocarcinoma of the prostate
* Testosterone < 50 ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy.
* Progressive disease after androgen deprivation.
* Patients who are receiving an antiandrogen as part of primary androgen ablation must demonstrate disease progression following discontinuation of antiandrogen.
* Karnofsky Performance Status ≥ 60%.
* One prior taxane based chemotherapy for prostate cancer. No more than two prior systemic therapies. At least four weeks have lapsed since prior therapy.
* Patients may have had prior ketoconazole, aminoglutethimide or corticosteroids for treatment of progressive prostate cancer.
* Patients receiving any other hormonal therapy, including any dose of megestrol acetate (Megace), Proscar (finasteride), any herbal product known to decrease PSA levels (e.g., Saw Palmetto and PC-SPES), or any systemic corticosteroid must discontinue the agent for at least 4 weeks prior to enrollment. Progressive disease must be documented after discontinuation of the hormonal therapy.
* Patients on stable doses of bisphosphonates that show subsequent tumor progression may continue on this medication; however, patients are not allowed to initiate bisphosphonate therapy within one month prior to starting therapy or throughout the study.
* Liver function tests (ALT, AST) less than 1.5 x upper limit of normal (ULN). The bilirubin must be within normal limits.
* ANC >1500/µl, Platelet count > 100,00/µl, Creatinine <1.5 x ULN, Hemoglobin > 8 mg/dl
* Ejection fraction ≥45%.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2006-07; Primary Completion 2008-08 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of the combination of ketoconazole and mitoxantrone plus GM-CSF on time to clinical progression in patients with prostate cancer that has progressed on prior therapy. | restaged every 9 weeks

SECONDARY OUTCOMES:
To evaluate the objective response frequency of the combination of ketoconazole and mitoxantrone plus GM-CSF. | restaged every 9 weeks
To investigate the safety of ketoconazole and mitoxantrone given in combination with GM-CSF. | AE reporting as occurs

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Amato, DO, Principal Investigator — Baylor College of Medicine - Methodist Hospital
Locations (1):
- Baylor College of Medicine - Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No